CLINICAL TRIAL: NCT05049109
Title: Integrated Telehealth After Stroke Care
Acronym: iTASC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Columbia University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAT7278; KL2TR001874 (NIH)
Record Dates: First submitted 2021-09-03; First posted 2021-09-17 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Blood Pressure; Stroke, Ischemic; Stroke Hemorrhagic
Keywords: Post-stroke BP management; BP control
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group X (Experimental): Patients who have had stroke and high blood pressure will participate in 5 telehealth visits, which will take place over 3 months. In addition, remote BP monitoring will be given.
  Interventions: Behavioral: Integrated Telehealth After Stroke Care; Behavioral: Usual post-stroke follow-up care
- Group Y (Active Comparator): Patients who have had stroke and high blood pressure will participate in 3 visits with primary care and stroke practitioner.
  Interventions: Behavioral: Usual post-stroke follow-up care

INTERVENTIONS:
Behavioral: Integrated Telehealth After Stroke Care — • 3 week and 8 week follow up visits with pharmacy through telehealth
  Patients will provide home blood pressure monitoring kits at discharge for the first three months. The telemonitor that can send blood pressure readings, wirelessly or through telephone, to a secure server where study staff can look at the readings. Any blood pressure readings that are not within normal range will trigger an alert to be sent to study staff who will then follow up with the patient. A trained staff member will show the patient how to use the blood pressure monitor. Patients will be asked to take blood pressure at least 3 days per week and transmit the readings to study staff.
  Patients will also be asked to wear an activity monitor starting at 4 weeks.
  Other Names: iTASC
  Arms: Group X
Behavioral: Usual post-stroke follow-up care — * 1-2 weeks follow up visit with primary care.
  * 4-6 week and 12 week follow up visit with stroke practitioner
  * At the end of the study, patients will be asked questions regarding their experience with the telehealth visits, health, medication taking and quality of life
  Other Names: Standard of care practice

SUMMARY:
In this pilot trial, the investigator will compare early post-stroke BP management using an integrated Telehealth After Stroke Care (iTASC), to usual care with a primary outcome of BP control defined by the mean 24-hr blood pressure through remote monitoring at 3 months and survey patient reported outcomes.

As this is a preliminary trial with a small sample, estimates derived will be used to plan the subsequent larger confirmatory trial. Descriptive statistics will characterize the randomized patients completing surveys and outcome assessments. The study will evaluate the primary clinical outcome (BP <140/90 mmHg) 90 days post-discharge as a function of treatment and adjusted for from baseline BP. Change from baseline BP will also be assessed as an outcome. Change in activity level and duration, as well as trends in sedentary time will be compared between arms, and pre- and post-intervention with visual tailored infographics in the intervention arm. Moderating effects of demographics will also be evaluated. Decisions regarding the pursuit of a subsequent trial will use the primary outcome, and analysis of all other measures will be hypothesis generating.

DETAILED DESCRIPTION:
Hypertension is the single most modifiable risk factor for prevention of secondary stroke. However, blood pressure (BP) remains poorly controlled after a stroke in up to 55% of survivors. Uncontrolled hypertension is associated with lack of support, low level of independence, poor medication adherence and limited self-efficacy. These barriers are compounded following stroke with limited access to outpatient care. Sedentary behavior prevalence after stroke is high in both inpatient and community settings. Addressing physical activity may be a simple strategy to help counter growing health concerns during the pandemic from social restrictions.

Pre-COVID, the investigator created TASC (Telehealth After Stroke Care), an interdisciplinary telehealth clinic inclusive of primary care, pharmacy, and stroke specialists to address complex post-acute transitions of care and improve BP control. However, BP monitoring alone at best has a modest impact on medication adherence and health behaviors. As telehealth services expand during the pandemic, there is greater incentivization to devise interventions that utilize remote care to foster effective self-management.

Improving health behaviors through remote monitoring and patient tailored feedback in an integrated post-acute stroke care model has not been studied. Integrated TASC (iTASC) is a telehealth intervention inclusive of interdisciplinary care and remote technology including BP monitoring and tracked activity, supplemented by infographics tailored with the patient's own data, to enhance BP control and drive health behavior modification.

In this proof-of-concept trial, the investigator will compare early post-stroke BP management among post-acute stroke patients at discharge randomized to the iTASC intervention or usual care (primary care and stroke physician follow up without remote monitoring) with a primary outcome of BP control defined by the mean 24-hr BP at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* have had a stroke and have high blood pressure

Exclusion Criteria:

* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Mean 24-hr systolic blood pressure (SBP) through remote monitoring at 3 months | 3 Months
  A home blood pressure telemonitor will send blood pressure readings, wirelessly or through telephone, to a secure server where study staff can look at the readings. Patients will be asked to take blood pressure at least 3 days per week. The readings will be averaged to obtain the mean measurement.
Difference in systolic blood pressure (SBP) from baseline to 3 months | Baseline and 3 months
  A home blood pressure telemonitor will send blood pressure readings, wirelessly or through telephone, to a secure server where study staff can look at the readings. This is designed to measure the change in SBP from baseline to 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Syeda Imama A. Naqvi, MD, Principal Investigator — Assistant Professor of Neurology at the Columbia University
Locations (1):
- CUIMC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided